CLINICAL TRIAL: NCT05959005
Title: Progression of Early Atrophic Lesions in Age-related Macular Degeneration (AMD).
Brief Title: Progression of Early Atrophic Lesions
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Monika Fleckenstein, Professor, University of Utah
Other Study IDs: IRB_00143184; 1R01EY034965-01 (NIH)
Record Dates: First submitted 2023-07-15; First posted 2023-07-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Age-Related Macular Degeneration
Keywords: iRORA; cRORA; Geographic Atrophy; non-exudative
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early GA lesions: Non-interventional
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention.

SUMMARY:
Early atrophic age-related macular degeneration (AMD) represents an important time window in the course of so far untreatable atrophic AMD, as patients typically experience only some degree of visual dysfunction, while being at significant risk for marked further loss of vision. To allow the precise evaluation of upcoming therapeutic interventions, a better understanding of the manifestation and variable disease progression is needed. This project aims to investigate refined tools to detect and monitor early atrophic AMD more accurately, including the impact on visual dysfunction and quality of life.

DETAILED DESCRIPTION:
The investigators will focus on a previously largely under-explored but highly relevant time window in progression of age-related macular degeneration (AMD), i.e., 'early atrophic AMD'. We postulate that a therapeutic effect in early atrophic AMD would probably save a large proportion of patients from progressive visual function loss and that it seems more justifiable to risk interventions in this time window than in earlier AMD stages. Against this background, a comprehensive knowledge of the natural disease progression in this potential therapeutic margin is essential. We will implement innovative multimodal high-resolution retinal imaging, comprehensive functional testing, and assessment of vision-related quality of life (VRQoL) combined with standardized and exploratory analysis strategies in a prospective, longitudinal study. This will enable the investigators to characterize and quantify the microstructural changes and associated functional and VRQoL deficits in eyes with early atrophic lesions with unprecedented accuracy. Knowledge of the strongest risk factors for accelerated disease progression will allow identification of patients at highest risk for visual function loss. Moreover, the investigator's hypothesis on disease-stage specific risk-factors may guide selection of therapeutic targets that are particularly susceptible in early atrophic AMD. Tailoring therapeutics to specific phenotypes and disease stages may be key to prevent irreversible vision loss and the associated reduced quality of life in patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 50 years and older of all ethnicities.
* Prior participation in the University of Utah IRB #00010201, "Genetic and Molecular Studies of Eye Disease" with written permission to be contacted for further clinical studies.
* Specifically, subjects must carry one or two risk alleles (subjects' nucleotides must be CC or CT to meet eligibility) at the CFH rs1061170 variant (CFH Y402H) or one or two risk alleles (subjects' nucleotides must be GT or TT to meet eligibility) at the ARMS2/HTRA1 rs10490924 variant. This genetic information will be available through the University of Utah IRB #00010201, "Genetic and Molecular Studies of Eye Disease".
* Study eye with at least one early atrophic lesion defined as:
* incomplete retinal pigment epithelium (RPE) and outer retinal atrophy (iRORA) (region of signal hypertransmission into the choroid, corresponding zone of attenuation or disruption of the RPE, and evidence of overlying photoreceptor degeneration that is, subsidence of the inner nuclear layer (INL) and outer plexiform layer (OPL), presence of a hyporeflective wedge in the Henle fiber layer (HFL), thinning of the outer nuclear layer (ONL), disruption of the external limiting membrane (ELM), or disintegrity of the ellipsoid zone (EZ), or
* complete RPE and outer retinal atrophy (cRORA) (homogeneous choroidal hypertransmission, absence of the RPE band measuring > 250µm, evidence of overlying photoreceptor degeneration) and total lesions size =< ½ disc area (DA) (corresponding to 1.27mm2 area) of all atrophic lesions measured on fundus-autofluorescence (FAF) imaging in the study eye.
* Sufficiently clear ocular media, adequate pupillary dilatation, and adequate fixation to permit quality fundus imaging and unbiased functional testing incl. fundus-controlled perimetry (FCP) testing.
* Ability to comply with study protocol timelines.

Exclusion Criteria:

* Signs or exudation defined as serous detachment of the sensory retina, intraretinal cystoid fluid, or subretinal/retinal hemorrhage in the study eye.
* cRORA lesion >1/2 disc area in the study eye at baseline.
* Any history of treatment of exudative macular neovascularization (MNV) in the study eye (e.g. type 1, type 2, mixed, polypoidal choroidal vasculopathy, and retinal angiomatous proliferation); Note: Non-exudative type 1 MNV in the study eye is NOT an exclusion criterion; non-exudative or exudative MNV in the fellow eye is not an exclusion criterion. Fellow-eyes may receive treatment of exudative MNV as part of clinical care.
* Any disease/disorder other than AMD in the study eye at the time of inclusion (e.g. monogenic retinal diseases, diabetic retinopathy, retinal detachment, previous retinal surgeries, myopic degeneration), uncontrolled glaucoma with intraocular pressure (IOP) of >30 mmHg (despite current pharmacological or non-pharmacological treatment) and uveitis.
* History of central retinal laser treatment, including photodynamic therapy (PDT) and subthreshold laser treatment for AMD in the study eye.
* Cataract surgery in the study eye within the last three months prior to enrollment. Laser-capsulotomy in the study eye within the last 2 weeks prior to enrollment.
* Current or previous participation in clinical trials investigating drugs or supplements in AMD (except vitamins and minerals).
* Current or previous participation (<3 months from termination of participation) in clinical trials investigating drugs or supplements in diseases other than AMD.
* Any concurrent ocular condition in the study eye (e.g. cataracts) that, in the opinion of the investigator, requires medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition or - if allowed to progress untreated - could likely contribute to loss of at least two Snellen equivalent lines of best-corrected visual acuity during the study period.
* Concomitant diseases that in the opinion of the investigator would make adherence to the examination schedule difficult or unlikely (e.g. personality disorder, chronic alcoholism, Alzheimer's Disease, drug abuse).
* Evidence of significantly uncontrolled concomitant diseases at the discretion of the investigator (e.g. cardiovascular, neurological, pulmonary, renal, hepatic, endocrine gastrointestinal disorder).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early atrophic lesions secondary to AMD in at least one eye.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in geographic atrophy (GA) lesion size | At months 36 from baseline
  Total GA lesion size will be determined by applying the RegionFinder® software on fundus-autofluorescence (FAF) with the aid of near-infrared (NIR) and optical coherence tomography ( OCT) images for the decision for the actual presence of early atrophic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fleckenstein, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided